CLINICAL TRIAL: NCT06868173
Title: Evaluation of the Analgesic Efficacy of Trigger Point Electroacupuncture in Patients With Chronic Low Back Pain: a Blinded Randomised Controlled Trial
Brief Title: Trigger Point Electroacupuncture Treatment in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Bui Pham Minh Man, Doctor of Philosophy, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2588/DHYD-HDDD
Record Dates: First submitted 2025-03-02; First posted 2025-03-10 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Chronic Low Back Pain (CLBP); Trigger Points
Keywords: Electro-acupuncture; Trigger points; Low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: A blinded randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The study participants will not know which electroacupuncture group they are in.
  The acupuncturist and the data processor are 2 different people.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electro-acupuncture at traditional points (Sham Comparator): 30 patients with non-radiating low back pain for at least three months and normal neurological examination received treatment electro-cupuncture at traditional points for 10 sessions over 4 weeks, electroacupuncture was administered once per session, three sessions per week, on alternate days, with rest on Saturdays and Sundays. Visual analogue scale (VAS) will be recorded after 1 session, 3 session, 5 session, 7 session and 10 session. BPI index and Trigger point count will be recorded after 1 session, 5 session, 10 session.
  Interventions: Device: Electro-acupuncture
- Electro-acupuncture at the Trigger point (Active Comparator): 30 patients with non-radiating low back pain for at least three months and normal neurological examination received treatment electro-acupuncture at the Trigger point for 10 sessions over 4 weeks, electroacupuncture was administered once per session, three sessions per week, on alternate days, with rest on Saturdays and Sundays. Visual analogue scale (VAS) will be recorded after 1 session, 3 session, 5 session, 7 session and 10 session. BPI index and Trigger point count will be recorded after 1 session, 5 session, 10 session.
  Interventions: Device: Electro-acupuncture

INTERVENTIONS:
Device: Electro-acupuncture — Electroacupuncture at Trigger Points is electroacupuncture at predetermined trigger points. Electroacupuncture at traditional acupoints is electroacupuncture at the following points: Jiaji (L2-L5), Yaoyangguan (GV3), Shendu (BL23), Dachangdu (BL25), and Weizhong (BL40).

SUMMARY:
Electroacupuncture is an application of acupuncture combined with electrical stimulation of acupuncture points through acupuncture needles to achieve faster pain relief than acupuncture. Recently, research has shown that Trigger point acupuncture has a significant effect in reducing pain better than acupuncture on acupoints in patients with chronic low back pain. However, no research has compared the pain relief effect between Trigger Point electroacupuncture and electroacupuncture on acupoints in patients with chronic low back pain. This study was conducted to address this question.

DETAILED DESCRIPTION:
Participants and Methods: A blinded randomized controlled clinical trial was conducted involving 60 chronic low back pain participants, randomly divided into two groups (A and B): 30 receiving electroacupuncture at the Trigger point (group A) and 30 receiving electroacupuncture on the meridian (group B) for 10 sessions. The primary outcomes were visual analogue scale (VAS), BPI index, and Trigger point count.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 or older who consented to participate in the study;
* Individuals experiencing LBP persisting for more than 3 months with an average VAS score of 5 cm or over;
* Patients displaying trigger points in back

Exclusion Criteria:

* Major trauma or systemic disease such as rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, Scheuermann disease;
* Systemic symptoms such as weight loss, fever of unknown origin, anorexia, personal history of malignancy, diffuse pain and joint stiffness;
* Symptoms of infection such as fever, meningeal irritation signs, photophobia;
* Symptoms of central motor neuron damage such as Hoffmann sign, Babinski sign, hyperreflexia, spasticity, incontinence, sexual dysfunction;
* Symptoms of serious acute diseases such as myocardial infarction (chest pain, sweating, shortness of breath), arterial dissections (tearing sensation, headache, blurred vision);
* Conditions unsuitable for acupuncture such as inflammation of skin in need of acupuncture, weak or exhausted patients, severe comorbidities;
* Being treated with other methods. Elimination criteria: Patients experiencing adverse events from the intervention leading to their discomfort and withdrawal from the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Comparison of VAS pain intensity between electroacupuncture at the trigger point and electroacupuncture traditional point group | Baseline, after 3 sessions, after 5 sessions, after 7 sessions, after 10 sessions
  With the VAS, participants were asked to make a hatch mark on a 100 mm line that represents their average pain intensity. These were then converted to a numerical score for each face (i.e. 0, 2, 4, 6, 8, or 10), depending on the face selected. The end-point descriptors for VAS was "No pain" (0, 0 mm, and the face representing no pain, respectively) and "The most intense pain imaginable" (10, 100 mm, and the face representing the most intense pain level, respectively).

SECONDARY OUTCOMES:
Comparison of BPI index between electroacupuncture at the trigger point and electroacupuncture traditional point group. | Baseline, after 5 sessions, and after 10 sessions
  The BPI gives two main scores: a pain severity score and a pain interference score. The pain severity score is calculated from the four items about pain intensity. Each item is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score, ranging from 0 to 40. The pain interference score corresponds to the item on pain interference. The seven sub-items (general activity, mood, walking ability, normal walk, relations with other people, sleep, and enjoyment of life) are rated from 0, does not interfere, to 10, completely interferes, and contributes with the same weight to the final score, ranging from 0 to 70. The first item, pain drawing diagrams (painful and most painful areas) and the items on pain relief treatment or medication (list of the treatments and amount of relief) do not contribute to the scoring. It takes approximately 5 minutes to complete the BPI.

OTHER OUTCOMES:
Comparison of trigger point count between electroacupuncture at the trigger point and electroacupuncture traditional point group | Baseline, after 5 sessions, and after 10 sessions
  Determine the number of trigger points at each survey time.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medical Center HCMC - Branch no.3, Ho Chi Minh, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Leite PMS, Mendonca ARC, Maciel LYS, Poderoso-Neto ML, Araujo CCA, Gois HCJ, Souza JHS, DeSantana JM. Does Electroacupuncture Treatment Reduce Pain and Change Quantitative Sensory Testing Responses in Patients with Chronic Nonspecific Low Back Pain? A Randomized Controlled Clinical Trial. Evid Based Complement Alternat Med. 2018 Oct 8;2018:8586746. doi: 10.1155/2018/8586746. eCollection 2018. PMID 30402136
- [Background] Schliessbach J, van der Klift E, Arendt-Nielsen L, Curatolo M, Streitberger K. The effect of brief electrical and manual acupuncture stimulation on mechanical experimental pain. Pain Med. 2011 Feb;12(2):268-75. doi: 10.1111/j.1526-4637.2010.01051.x. Epub 2011 Jan 28. PMID 21276188
- [Background] Itoh K, Katsumi Y, Kitakoji H. Trigger point acupuncture treatment of chronic low back pain in elderly patients--a blinded RCT. Acupunct Med. 2004 Dec;22(4):170-7. doi: 10.1136/aim.22.4.170. PMID 15628774
- [Background] Itoh K, Katsumi Y, Hirota S, Kitakoji H. Effects of trigger point acupuncture on chronic low back pain in elderly patients--a sham-controlled randomised trial. Acupunct Med. 2006 Mar;24(1):5-12. doi: 10.1136/aim.24.1.5. PMID 16618043